CLINICAL TRIAL: NCT03324607
Title: Effects of Glycopyrrolate/Formoterol (Bevespi) on Ventilation and Gas Exchange Abnormalities in COPD Assessed by 129Xe MRI
Brief Title: Effects of Bevespi on Ventilation and Gas Exchange Abnormalities in COPD Assessed by 129Xe MRI
Acronym: COPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00086693
Record Dates: First submitted 2017-09-29; First posted 2017-10-27 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): glycopyrrolate/formoterol (Bevespi) 2 puffs twice a day taken for two weeks, started after completion of the study XeMRI. A follow up xeMRI occurs at the end of the two weeks of taking the Bevespi in a Pre-post study design.
  Interventions: Drug: hyperpolarized 129Xe gas MRI; Drug: Bevespi Aerosphere

INTERVENTIONS:
Drug: hyperpolarized 129Xe gas MRI — There will be MRI imaging before the treatment with Bevespi and another one 2 weeks after use Bevespi. Images obtained using 129Xe MRI will be compared with standard lung function tests that are used routinely in the clinic, 6 minute walk test that assesses walking ability and several questionnaires that assess shortness of breath and life quality.
  Other Names: 129Xe MRI
Drug: Bevespi Aerosphere — There will be MRI imaging before the treatment with Bevespi and another one 2 weeks after use Bevespi.
  Other Names: Inhaler

SUMMARY:
The purpose of this study is to determine whether the new inhaler, Bevespi improves lung function. Magnetic resonance imaging (MRI) using inhaled hyperpolarized 129Xe gas, that can provide useful images of the functioning of the lung will be used as a new measure to determine change in function. The investigator anticipate these images will provide more specific information about lung disease than standard lung function tests in response to treatment.

DETAILED DESCRIPTION:
The study will characterize ventilation and gas transfer distributions in GOLD II and III COPD patients and assess the potential for these physiological parameters as a novel phenotyping method using Magnetic resonance imaging (MRI) using inhaled hyperpolarized 129Xe gas.

The study will additionally quantify regional ventilation and gas transfer response to glycopyrrolate/formoterol in GOLD II and III COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by post-bronchodilator spirometry demonstrating (forced expiratory volume at 1 second(FEV1)/forced vital capacity (FVC) < 0.70 and forced expiratory volume at 1 second (FEV1) in GOLD 2 or 3 stage (30%≤ (forced expiratory volume at 1 second [FEV1] < 80%)
* Willing and able to give informed consent and adhere to visit/protocol schedules
* Women of childbearing potential must have a negative urine pregnancy test

Exclusion Criteria:

* Upper respiratory tract infection within 6 weeks
* Chronic systemic corticosteroid use > 10 mg/day of prednisone

  * Chronic oxygen use (intermittent or continuous)
  * Previous lung resection surgery or decortication
  * Previous history of pneumothorax
  * Evidence of interstitial, occupational or chronic infectious lung disease by imaging studies
  * History of exposure to occupational or environmental hazards that are known to cause lung diseases
  * For women of child bearing potential, positive pregnancy test
  * Major chronic illnesses which in the judgement of the study physician would interfere with participation in the study
  * Patients who are not willing to withhold COPD inhalers for the run-in period.

    * MRI is contraindicated based on responses to MRI screening questionnaire
    * Subject is pregnant or lactating
    * Respiratory illness of a bacterial or viral etiology within 30 days of MRI
    * Subject has any form of known cardiac arrhythmia
    * Subject does not fit into 129Xe vest coil used for MRI
    * Subject cannot hold his/her breath for 15 seconds
    * Subject deemed unlikely to be able to comply with instructions during imaging

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuh Chin Huang, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma, Allergy, and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2018 and October 2019, 52 outpatient pulmonary clinic patients were approached about potential participation in the study. Twenty-six participants signed a written informed consent prior to enrollment and the HIPAA-compliant study protocol was approved by the Institutional Review Board of Duke University Medical Center (Pro00086693). Six participants were either withdrawn by the PI or voluntarily withdrew prior to starting the study.
Pre-assignment Details: All subjects who were on regular inhalation therapies for COPD underwent a wash-out period of 7-14 days, during which time they stopped all inhaled corticosteroids, long-acting beta agonist (LABA), and long-acting muscarinic receptor antagonist (LAMA). The subjects were allowed to use inhaled albuterol as needed.
Groups:
- Treatment: Twenty patients with a pulmonologist's diagnosis of either GOLD II or III COPD and no significant comorbidities were recruited. One patient was excluded from data analysis due to poor image signal-to-noise ratio, and two patients did not have both pre- and post-treatment ventilation images; thus, a total of 17 patients (8M; 9F) were included in the data analysis. The mean age was 64.3 ± 4.9.
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects who were on regular inhalation therapies for COPD underwent a wash-out period of 7-14 days, during which time they stopped all inhaled corticosteroids, long-acting beta agonist (LABA), and long-acting muscarinic receptor antagonist (LAMA). The subjects were allowed to use inhaled albuterol as needed.
Groups:
- Treatment: Twenty subjects completed the study. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit; thus, a total of 17 subjects (8M 9F) were included in the data analysis. Subjects were treated with Bevespi 2 puffs twice a day for 2 weeks.
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Age measured in years Population: 3 subjects were excluded due to incomplete data or poor data quality
  years
    number analyzed (Participants) | 17
    (all) | 64 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 subjects were excluded due to incomplete data or poor data quality
  Participants
    number analyzed (Participants) | 17
    Female | 9
    Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0
  Non-Hispanic | 17
  Caucasian | 17
  African-American | 0

OUTCOME MEASURES:

1. Primary Outcome: Ventilation Distribution as Measured by Ventilation Defect+Low Percent
Description: The ventilation distribution as measured by ventilation defect+low percent is to measure the area of the lung that has no air.
Time Frame: Week 2
Population: 17 participants were included in the data analysis. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
Measure: Mean (Standard Deviation); unit: percentage of total ventilation
Groups:
- Treatment: glycopyrrolate/formoterol (Bevespi) 2 puffs twice a day taken for two weeks, started after completion of the study XeMRI. A follow up XeMRI occurs at the end of the two weeks of taking the Bevespi in a Pre-post study design.
  hyperpolarized 129Xe gas MRI: There will be MRI imaging before the treatment with Bevespi and another one 2 weeks after use Bevespi. Images obtained using 129Xe MRI will be compared with standard lung function tests that are used routinely in the clinic, 6 minute walk test that assesses walking ability and several questionnaires that assess shortness of breath and life quality.
  Bevespi Aerosphere: There will be MRI imaging before the treatment with Bevespi and another one 2 weeks after use Bevespi.
Arm/Group | Treatment
Number analyzed (Participants) | 17
percentage of total ventilation
  Baseline | 57.8 (8.4)
  Week 2 | 52.5 (10.6)
Statistical Analysis 1: Comparison: Treatment; Test type: Other; p = 0.006, Paired t-test

2. Primary Outcome: Barrier Uptake.
Description: Diffusion of Xe gas across the lung membrane into the blood. This measures how well oxygen goes through the lung into the blood.
Time Frame: 2 weeks
Population: 17 patients with GOLD 2 or 3 COPD 17 participants were included in the data analysis. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 17
Participants
  increase in barrier uptake | 13
  No increase in barrier uptake | 4

3. Primary Outcome: Red Blood Cell (RBC) Uptake
Description: Amount of Xe gas that enters the blood stream after it diffuses across the lung membrane
Time Frame: 2 weeks
Population: GOLD 2 and 3 COPD 17 participants were included in the data analysis. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 17
Participants
  Decrease in red blood cell (RBC) uptake | 10
  No decrease in red blood cell (RBC) uptake | 7

4. Secondary Outcome: Pulmonary Function Test - Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible, as measured by spirometry.
Time Frame: 2 weeks
Population: One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
  17 participants were included in the data analysis. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment
Number analyzed (Participants) | 17
ml | 342 (286)

5. Secondary Outcome: Pulmonary Function Test - Forced Expiratory Volume-one Second (FEV1)
Description: FEV1 is a lung airflow measure to assess the amount of air that can be blown out in one second.
Time Frame: 2 weeks
Population: One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment
Number analyzed (Participants) | 17
ml | 219 (168)

6. Secondary Outcome: Pulmonary Function Test - Total Lung Capacity (TLC)
Description: Total Lung Capacity (TLC) is the volume in the lungs at a maximal inhalation.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment
Number analyzed (Participants) | 17
ml | 183 (411)

7. Secondary Outcome: Pulmonary Function Test - Residual Volume (RV)
Description: Residual volume (RV) is the volume of air remaining in the lungs after a maximal exhalation.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment
Number analyzed (Participants) | 17
ml | -108 (508)

8. Secondary Outcome: Pulmonary Function Test - Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: DLCO measures the ability of oxygen to travel from the air sacs of the lungs to the blood stream.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Treatment
Number analyzed (Participants) | 17
mL/min/mmHg | 0.2 (1.3)

9. Secondary Outcome: 6-minute Walk Test (6MWT)
Description: The 6-minute walk test (6MWT) measures the distance walked at a natural pace for 6 minutes.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment
Number analyzed (Participants) | 17
meters | 16.2 (37.6)

10. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Score
Description: The SGRQ is used to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 17
score on a scale | -1.2 (5.8)

11. Secondary Outcome: Rating of Perceived Dyspnea (RPD) Scale
Description: A patient reported outcome to measure perceived exertion during physical activity. The RPD scale goes from 0 to 10, where 0 = no shortness of breath at all and 10 = maximal shortness of breath (needing to stop the exercise or activity).
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 17
score on a scale | -0.75 (2.33)

12. Secondary Outcome: COPD Assessment Test (CAT) Score
Description: Functional measurement for COPD patients. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 17
score on a scale | -3.8 (4.5)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
20 subjects completed the study. One subject was excluded from data analysis due to poor image signal-to-noise ratio (SNR), and two elected not to return for a post-treatment visit; thus, a total of 17 subjects (8M 9F) were included in the data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03324607/Prot_SAP_000.pdf